CLINICAL TRIAL: NCT06699667
Title: CT Findings in Surgically Treated Focal Pancreatic Disease- A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas S Kristensen, Associate Professor, Chief Physician, Rigshospitalet, Denmark
Other Study IDs: RH -2015-07, 03616
Record Dates: First submitted 2024-11-14; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Pancreatitis
Keywords: autoimmune pancreatitis; pancreatic ductal adenocarcinoma; radiology
MeSH Terms: conditions — Autoimmune Pancreatitis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed tomography

SUMMARY:
To retrospectively investigate CT imaging features of autoimmune and chronic pancreatitis (AIP and CP) mimicking pancreatic ductal adenocarcinoma in surgically resected patients.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of autoimmune pancreatits or adenocarcinoma

Exclusion Criteria:

* No surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population in Copenhagen
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Imaging features of autoimmune pancreatitis | Time frame for each study object is the time between tumor board conference and surgery - typically 2-4 weeks
  Patients with a final histopathological diagnosis of autoimmune pancreatitis is identified from pancreatic surgery database and compared with matched control groups. Imaging features available at the primary tumor board conference are evaluated blinded to the final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Carsten P Hansen, MD, Principal Investigator — Department of Surgery and Transplantation, Rigshospitalet

IPD SHARING:
Plan to Share IPD: Undecided